CLINICAL TRIAL: NCT05564325
Title: Real-time Deflectable Guidewire in Neuro-interventions Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artiria Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-01
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Unruptured Cerebral Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SmartGUIDE (deflectable guidewire) (Experimental)
  Interventions: Device: SmartGUIDE (deflectable guidewire)
- Standard of care guidewire (Active Comparator)
  Interventions: Device: Standard of care guidewire (different models may be used)

INTERVENTIONS:
Device: SmartGUIDE (deflectable guidewire) — SmartGUIDE is a deflectable guidewire for use in interventional procedures in the neurovasculature and the peripheral vasculature. It can be used to selectively introduce and position catheters and other interventional devices within the peripheral and neurovasculature. The device is a steerable guidewire with a deflectable tip. This allows adjusting the shape of the tip, dynamically, while the physician navigates the device in the patient's arterial and venous circulatory system.
  Arms: SmartGUIDE (deflectable guidewire)
Device: Standard of care guidewire (different models may be used) — The control device is any standard of care guidewire as per hospital routine indicated for neuro-interventional procedures.
  Arms: Standard of care guidewire

SUMMARY:
The aim of the study is to assess the safe and successful use of the SmartGUIDE guidewire in neuro interventions and to compare to standard of care guidewires on the market.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Informed consent signed by patient
* Confirmed cerebral unruptured aneurysm treatable via transcatheter approach

Exclusion Criteria:

* Pregnancy or lactation
* Known disorder of vascular fragility with propensity to vascular injury (e.g., Ehlers-Danlos syndrome)
* Known prior vascular stenosis or dissection or injury to vessels intended to be catheterized during study procedures
* Acute phase myocardial infarction or uncontrolled cardiac arrhythmia
* Uncontrolled serum electrolyte imbalance
* Bleeding disorder which limits the use of antiplatelet and/or anticoagulant therapy
* Known contraindication to intravascular contrast material that cannot be adequately controlled with pre-medication
* Known hypersensitivity to Nickel
* Subjects currently enrolled in another investigational device or drug study that clinically interferes with the current study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Performance | During index procedure
  Intra-procedural technical success defined as successful navigation of device to the vascular target vessel without need for shaping, removal or exchange.

SECONDARY OUTCOMES:
Usability | During index procedure
  Usability data (pushability, trackability, navigatability, shape retention, support, and proximal access complexity) collected through questionnaire completed by the physician. Measured through a Likert scale from 1-5.
Procedural times | During index procedure
  Procedural times (duration of tip reshaping, duration of access to target, duration of fluoroscopic exposition).
Safety - intra- and postprocedural | During index procedure and up to 48 hours post procedure
  Adverse events, measured by the occurrence of adverse events
Device Deficiencies | During index procedure
  Intraprocedural device deficiencies, measured by the occurrence of device deficiencies/malfunctions

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Machi, Professor, Principal Investigator — Geneva University Hospital - HUG
Locations (2):
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland
  - Geneva University Hospital - HUG, Geneva

IPD SHARING:
Plan to Share IPD: No